CLINICAL TRIAL: NCT07087158
Title: A Multicenter, Randomized, Open-Label, Active-Controlled Phase II Study Evaluating the Efficacy and Safety of IBR854 Combined With Pazopanib Versus Pazopanib in Advanced Renal Cell Carcinoma
Brief Title: A Study of IBR854 Combined With Pazopanib Versus Pazopanib in Advanced Renal Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imbioray (Hangzhou) Biomedicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBR854-203
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: IBR854
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): IBR854 + Pazopanib
  Interventions: Drug: IBR854; Drug: Pazopanib
- Control arm (Active Comparator): Pazopanib
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: IBR854 — Every 21 days is one cycle, and IBR854 will be dosed in a route of intravenous infusion on day 1 and day 8 of each cycle with a fixed dose of 9.0×10^9 cells.
  Arms: Experimental arm
Drug: Pazopanib — Pazopanib will be dosed orally once daily without food (at least 1 hour before or 2 hours after a meal) with a fixed dose of 800mg.

SUMMARY:
This is a multicenter, randomized, open-label, active-controlled Phase II clinical study evaluating the efficacy and safety of IBR854 combined with Pazopanib versus Pazopanib in Advanced Renal Cell Carcinoma.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, active-controlled study. Eligible patients with Advanced Renal Cell Carcinoma who meet all inclusion criteria and none of the exclusion criteria will be randomly assigned in a 2:1 ratio to either the experimental arm or the control arm.

* Experimental arm: IBR854 in combination with Pazopanib
* Control arm: Pazopanib The primary endpoint is PFS per RECIST 1.1. Efficacy and safety datas will be continuously collected until criteria for discontinuation are met.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years old
2. Advanced clear cell renal cell carcinoma confirmed by histology or cytology and not amenable to curative surgery.
3. Has not received any previous systemic anti-tumor treatment for advanced renal cell carcinoma.
4. Expected survival period is at least 3 months.
5. ECOG performance status of 0 or 1, or KPS score of at least 70.
6. Has measurable disease per RECIST 1.1.
7. Organ function should meet the following criteria:

   1. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L; Platelet (PLT) ≥90×10^9/L; Hemoglobin (Hb) ≥ 90 g/L (no blood transfusion or hematopoietic stimulator treatment within 7 days).
   2. Albumin ≥ 30 g/L; Total bilirubin ≤1.5×ULN (for subjects with Gilbert's syndrome, it can be ≤3×ULN); ALT and AST ≤1.5×ULN (If liver metastasis is combined, ALT and AST≤3×ULN).
   3. Creatinine (Cr) ≤1.5 × ULN; Creatinine clearance (Ccr) (to be calculated only when Cr > 1.5× ULN) > 50 ml/min (Cockcroft-Gault formula).
   4. Activated partial thrombin time (APTT) ≤1.5×ULN, International normalized ratio (INR) ≤1.5×ULN.
8. Voluntarily sign the informed consent form, understand the study and be willing to follow the protocol and complete all experimental procedures.

Exclusion Criteria:

1. Documented central nervous system metastases.
2. Received prior antineoplastic therapy (including chemotherapy, biologic therapy, immunotherapy, or Chinese traditional medicines with antitumor indications) before the first dose of study treatment.
3. Has received major surgery (grade 3 or 4 as defined in the Measures for the Administration of Clinical Application of Medical Technology) within 28 days before the first dose of study treatment and has not yet recovered from which; or any planned curative surgery for renal cell carcinoma during the study.
4. History of another malignancy within 5 years before the first dose of study treatment, except for Lung carcinoma in situ, low-risk early-stage prostate cancer, or cured basal-cell carcinoma, squamous-cell carcinoma of the skin, cervical carcinoma in situ, or papillary thyroid carcinoma.
5. Clinically significant gastrointestinal abnormalities such as malabsorption syndrome, major gastric or small-bowel resection that may affect drug absorption, active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other conditions increasing the risk of perforation; or history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days before the first dose of study treatment.
6. Systemic corticosteroids (>10 mg/day prednisone or equivalent) or other immunosuppressive agents required within 2 weeks before the first dose or anticipated during study treatment, except for:

   1. Topical, intranasal, or inhaled corticosteroids.
   2. Corticosteroids as premedication for infusion-related or hypersensitivity reactions (e.g., premedication for CT imaging).
   3. Replacement therapy such as levothyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency.
   4. Low-dose corticosteroids for orthostatic hypotension.
7. Clinically significant cardiovascular or cerebrovascular disease documented by any of the following:

   1. Ischemic stroke (excluding silent lacunar infarction) or severe thromboembolic event within 6 months before the first dose of study treatment.
   2. Myocardial infarction, unstable angina, congestive heart failure, or clinically significant arrhythmia within 6 months before the first dose of study treatment.
   3. New York Heart Association (NYHA) class ≥ II heart failure before the first dose of study treatment.
   4. QTcF interval >450 ms (men) or >470 ms (women) before the first dose of study treatment.
   5. Left-ventricular ejection fraction (LVEF) ≤50 % before the first dose of study treatment.
8. Prior organ transplant, except corneal transplant; prior allogeneic stem-cell transplant.
9. Hepatitis B surface antigen (HBsAg) positive with HBV DNA >500 IU/mL or >2,500 copies/mL, or hepatitis C antibody positive with detectable HCV RNA, or known HIV infection, or active tuberculosis.
10. Interstitial lung disease or non-infectious pneumonitis that is currently symptomatic or has previously required systemic corticosteroids, in the opinion of the investigator likely to interfere with toxicity assessment or management.
11. Any severe, progressive, or uncontrolled medical condition that, in the investigator's judgment, makes the subject unsuitable for the study, including but not limited to:

    1. Infection requiring systemic therapy.
    2. Symptomatic pleural, pericardial, or ascitic fluid requiring or having undergone drainage within 2 weeks before the first dose (minimal asymptomatic effusion, third-spacing due to hypoalbuminaemia, or cases where benefit outweighs risk may be allowed).
    3. History of coagulopathy (e.g., deep-vein thrombosis) or severe bleeding diathesis; clinically significant bleeding event (e.g., gastrointestinal bleeding) within 1 month before the first dose.
    4. History of severe psychiatric disorder.
    5. Any other condition that, in the investigator's opinion, renders study participation riskier than beneficial.
12. Prior grade 3-4 immune-related adverse events that, in the investigator's judgment, should be excluded.
13. Severe allergic or hypersensitivity disorders, significant drug allergies (including to investigational agents), or known hypersensitivity to any component of the study drug, including severe reactions to monoclonal antibodies.
14. Participation in another clinical trial and receipt of an investigational agent within 28 days before the first dose of study treatment.
15. Clinically significant organ dysfunction or comorbidity likely to interfere with protocol adherence.
16. Live vaccine received within 30 days before the first dose, or planned during the study or within 1 month after the last dose.
17. Pregnant or breast-feeding women (women who agree to discontinue breast-feeding before signing informed consent may be enrolled).
18. Any other condition or circumstance that, in the investigator's opinion, unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Approximately 2 years
  The time from randomization to the first radiologically confirmed disease progression or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 4 years
  The time from randomization to death from any cause (whichever occurs first).
Objective Response Rate (ORR) | Approximately 2 years
  Proportion of participants who have a CR or PR per RECIST 1.1.
Disease Control Rate (DCR) | Approximately 2 years
  Proportion of participants who have a CR, PR or SD per RECIST 1.1.
Duration of Response (DoR) | Approximately 2 years
  The time from the date of first response until date of the first radiologically confirmed disease progression per RECIST 1.1.
Adverse Events (AEs) | Approximately 2 years
  The incidence and severity of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- The Cancer Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No